CLINICAL TRIAL: NCT03747159
Title: A Randomized Trial to Investigate the Reset of Humoral Autoimmunity by Combining Belimumab with Rituximab in Severe Systemic Lupus Erythematosus
Brief Title: Synergetic B-cell Immunomodulation in SLE - 2nd Study.
Acronym: SynBioSe-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Dutch Kidney Foundation (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Y.K.Onno Teng, Dr. Y.K.O. Teng, Nephrologist, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL65720.058.18
Record Dates: First submitted 2018-10-12; First posted 2018-11-20 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: systemic lupus erythematosus; lupus nephritis; systemic autoimmune disease; glomerulonephritis; autoimmune glomerulonephritis; membranoproliferative glomerulonephritis; renal insufficiency; renal failure
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis; Glomerulonephritis; Glomerulonephritis, Membranoproliferative; Renal Insufficiency | interventions — belimumab

STUDY DESIGN:
Intervention Model Description: Multi-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BLM+RTX treatment arm (Experimental): Intervention 1 Belimumab injection: subcutaneous weekly injections with 200mg belimumab (BML) for the duration of the entire study period of two years.
  Intervention 2 Rituximab infusion: Two intravenously infusions of 1000mg rituximab (RTX) at week 4 and week 6 after the start of belimumab.
  Intervention 3: Standard of care: induction therapy with three intravenously infusions methylprednisolone of 1000mg (or 500mg if weight is below 60kg), oral prednisolone 60mg with a quick tapering scheme to reach 5mg in 10 weeks and mycofenolate mofetil start dosis 500mg twice daily with maximum dosis of 2000mg twice daily depending on tolerance and area under curve (AUC) aimed at 60mg*hour/L.
  Interventions: Drug: Belimumab Injection
- Standard of Care treatment arm (No Intervention): Intervention 1: Standard of care: induction therapy with three intravenously infusions methylprednisolone of 1000mg (or 500mg if weight is below 60kg), oral prednisolone 60mg with a quick tapering scheme to reach 5mg in 10 weeks and mycofenolate mofetil start dosis 500mg twice daily with maximum dosis of 2000mg twice daily depending on tolerance and area under curve (AUC) aimed at 60mg*hour/L.
  Optional intervention: (if patients flare or are non-responders on mycofenolate mofetil + prednisolone) : Two intravenously infusions of 1000mg rituximab at week 4 and week 6 after the start of belimumab.

INTERVENTIONS:
Drug: Belimumab Injection — Weekly injection of belimumab prior to two infusions of rituximab with continuation of the belimumab as maintenance therapy
  Other Names: Benlysta subcutaneous injection of 200mg
  Arms: BLM+RTX treatment arm

SUMMARY:
In follow-up of the previous SynBioSe Study the present study is a randomized controlled trial designed to further investigate the long-term clinical and imunological efficacy of combination B-cell targeting by starting treatment with belimumab (anti-BAFF) followed by rituximab(anti-CD20) in lupus nephritis patients.

DETAILED DESCRIPTION:
Rationale:

The SynBioSe-1 study is the first study to comprehensively describe the clinical and immunological effects of combining rituximab (RTX) and belimumab (BLM) in patients with systemic lupus erythematosus (SLE). From the pioneering SynBioSe-1 study, we have learned that combining RTX+BLM was safe and well-tolerated with important clinical responses. Immunologically, we unexpectedly observed that long-term B-cell depletion was not achieved due to migration of mature B-cells triggered by depletion of BAFF serum levels. The latter observation was in contrast to the study's null-hypothesis that combination therapy would lead to long-term B-cell depletion. The contrary was demonstrated, namely the relative early recirculation of mature B-cells. As such, the immunological and clinical lessons from the SynBioSe-1 study in conjunction with accumulating data from several large studies on combination B-cell targeted treatment have led to the postulation that starting treatment with RTX+BLM would result in an improved B-cell targeting strategy, notably on tissue-resident autoreactive B-cells, associated with improved long-term clinical disease amelioration. Therefore, the present SynBioSe-2 study is designed to further investigate the long-term clinical and imunological efficacy of combination B-cell targeting by starting treatment with belimumab followed by rituximab.

Objectives:

The primary objective is to assess whether combination treatment BLM+RTX will lead to reduced treatment failure and the improvement of pivotal, SLE-specific autoimmune phenomena compared to SLE patients treated with standard of care.

Study design:

a multi-center, randomized, controlled, open-label study

Study population:

SLE patients with a severe flare with major organ involvement or persistent high disease activity despite conventional treatment

Intervention:

In addition to standard therapy, SLE patients will receive self-administered, subcutaneous injections of belimumab every week for the entire study period and 2 infusions of rituximab 1000 mg on day 28 (week 4) and day 42 (week 6).

Main study parameters:

The primary clinical efficacy parameter is the treatment failure rate during the 2 years study period. Secondary endpoints are clinical and non-biased immunological effects of the treatment summarized as follows: reduction of disease relevant autoantibodies, in particular anti-dsDNA autoantibody production at 28 weeks, total renal response rate at 28 weeks, regression of immune complex-mediated excessive neutrophil extracellular traps (NET) formation at 28 weeks; sustained, long-term B-cell depletion during 104 weeks; sustained reduction of relevant anti-nuclear autoantibodies, including seroconversion during 104 weeks; and sustained regression of immune complex-mediated excessive neutrophil extracellular traps (NET) formation during 104 weeks. Additionally, the study will perform safety and toxicity monitoring according to Common toxicity Criteria (CTC) developed by the National Cancer Institute (NCI) with the use of Common Terminology Criteria for Adverse Events (CTCAE) and evaluate the reduction of concomitant immunosuppression and the number of moderate and severe flares during study follow-up.

Study duration: 104 weeks.

Nature and extent of the burden and risks associated with participation and potential benefits:

The study will include SLE patients with a severe flare necessitating remission induction treatment with intensive immunosuppression. The use of belimumab followed by rituximab can ameliorate disease activity even more than conventional treatment in the short-term and contribute to the successful tapering of concomitant immunosuppressive treatment. The latter will possibly lead to the reduction of infectious complication as compared to conventional treatment. The risks are predominantly related to the side effect profile of rituximab and belimumab and infectious complications of long-term B-cell depletion.

ELIGIBILITY:
Inclusion Criteria:

1. Have a clinical diagnosis of SLE according to the SLICC criteria 2012
2. Severe, active SLE disease defined as a situation in which 1 or more of the following criteria are met:

   1. SLEDAI-2K (SLE Disease Activity Index) with 12 or more points
   2. New or worse SLE-related activity of major organs, i.e.: CNS-SLE (includes NPSLE), vasculitis, nephritis, pericarditis and/or myocarditis, myositis, thrombocytopenia < 60, hemolytic anemia < 4.4mmol/L (=7.0g/dL)
   3. high disease activity that requires or warrants induction treatment by switching to or increasing dosage of oral mycophenolate
3. New, persisting or progressive disease activity despite the use of conventional maintenance immunosuppressive treatment (e.g. mycophenolate or azathioprine)
4. Positive for relevant SLE-specific autoantibodies defined as a situation in which 1 or more of the following criteria are met:

   1. ANA seropositivity, as defined by a positive ANA-titer ≥ 1:80, before and at screening :

      * Positive test results from 2 independent time points within the study screening period; OR
      * One positive historical test result and 1 positive result during the screening period. Historical documentation of a positive test of ANA (eg, ANA by HEp-2 titer, ANA by ELISA) must include the date of the test.
   2. Anti-DNA seropositivity, as defined by a positive anti-dsDNA serum antibody ≥ 30 IU/mL, before and at screening:

      * Positive test results from 2 independent time points within the study screening period.
      * One positive historical test result and 1 positive result during the screening period. Historical documentation of a positive test of anti-dsDNA (eg, anti-dsDNA by Farr assay or ELISA) must include the date of the test.
5. Female subjects are eligible to enter the study if she is:

   * Not pregnant or nursing
   * Of non-child-bearing potential (i.e. after hysterectomy, postmenopausal, bilateral ovariectomy or documented bilateral tubal ligation or other permanent female sterilization procedure)
   * in agreement to not become pregnant (if female subjects of childbearing potential) and therefore must be sexually inactive by abstinence or use contraceptive methods with a failure rate of < 1%.

Exclusion Criteria:

1. Active pregnancy, as proven by a positive urine beta-HCG test or a positive serum beta-HCG
2. Significant hypogammaglobulinemia (IgG < 4.0 g/L) or an IgA deficiency (IgA < 0.1 g/L)
3. Immunization with a live vaccine 1 month before screening
4. Active infection at time of screening, as follows:

   * Hospitalization for treatment of infection within previous 60 days of day 0 of the study
   * Use of parenteral (intravenous of intramuscular) antibiotics (including anti-bacterials, anti-virals, anti-fungals or anti-parasitic agents) within previous 60 days of day 0 of the study
   * Serological evidence of viral hepatitis defined as: patients positive for HbsAg test or HBcAb or a positive hepatitis C antibody not treated with antiviral medication
5. Have a historically positive HIV test or test positive at screening for HIV
6. Have a history of a primary immunodeficiency
7. Have a neutrophil count of < 1.5x10E9/L
8. Have a significant infection history that in the opinion of the investigator would make the candidate unsuitable for the study
9. Have a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies
10. Have any other clinically significant abnormal laboratory value in the opinion of the investigator
11. Have current drugs or alcohol abuse or dependence within 365 days prior to Day 0 of the study
12. Have an active malignant neoplasm or one in the history of the last 5 years, except basal cell or squamous cell carcinoma of the skin treated with local resection only or carcinoma in situ of the uterine cervix treated locally and with no evidence of metastatic disease for 3 years
13. Have evidence of serious suicide risk including any history of suicidal behavior in the last 6 months and/or any suicidal ideation in the last 2 months or who, in the investigator's opinion, poses a significant suicide risk
14. Have any other clinically significant abnormal laboratory value, any intercurrent significant medical or psychiatric illness that in the opinion of the investigator would make the candidate unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2026-06-07 (Estimated)

PRIMARY OUTCOMES:
Treatment failure rate | 2 years
  The treatment failure rate will be measured at 104 weeks in both treatment arms with the hypothesis that lower treatment failure rates will be obtained in the RTX+BLM arm.

SECONDARY OUTCOMES:
Change of disease relevant auto-antibodies present at baseline, in particular anti-dsDNA | 28 weeks
  All disease relevant auto-antibodies will be measured at 28 weeks and compared to baseline with the hypothesis that a better reduction will be obtained in the RTX+BLM arm.
Sustained change of autoantibody production | 2 years
  The sustained reduction of pathogenic autoantibodies, in particular anti-dsDNA autoantibodies
Seroconversion of disease relevant auto-antibodies | 2 years
  Seroconversion of pathogenic autoantibodies, in particular anti-dsDNA autoantibodies
Change of memory B-cell numbers | 28 weeks
  The detection of (autoreactive) memory B-cells by standardized flowcytometry and in B-cell culture assays
Sustained change of memory B-cell numbers | 2 years
  The detection of (autoreactive) memory B-cells by standardized flowcytometry and in B-cell culture assays
Change of immune complex-mediated excessive neutrophil extracellular traps (NET) formation | 28 weeks
  The quantification of ex vivo NET induction with a 3-dimensional, confocal microscopy technique
Sustained change of immune complex-mediated excessive neutrophil extracellular traps (NET) formation | 2 years
  The quantification of ex vivo NET induction with a 3-dimensional, confocal microscopy technique
Evaluation of the renal response | 2 years
  The number of partial and complete renal responders in case of lupus nephritis
Evaluation of the clinical response by SLEDAI | 2 years
  Patients will be monitored at frequent timepoints by the The Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K), with a minimum score of 0 and a maximum score of 105, with a higher score indicating a higher disease activity
Evaluation of the clinical response by SLICC | 2 years
  SLICC damage score (System Lupus International Collaborating Clinics/American College of Rheumatology Damage Index for Systemic Lupus Erythematosus) will be assesed at baseline, one year and two years, with a minimum score of 0 and a maximum score of 47, with a higher score indicating more damage
Evaluation of the clinical response by QoL questionnaires | 2 years
  QoL questionnaires will be assessed at multiple time points by the SF-36 (ShortForm-36) questionnaire, with a minimum score of 0 and a maximum score of 100, with a higher score indicating a higher quality of life
Evaluation of the clinical response by the amount of moderate and severe flares. | 2 years
  Patients will be monitored at frequent timepoints
Evaluation of the clinical response by the ability to reduce concomitant immunosuppression without flares | 2 years
  Patients will be monitored at frequent timepoints
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 2 years
  Patients will be monitored at frequent timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Y.K.O. Teng, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (4):
- Netherlands (4):
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Radboud University Medical Center, Nijmegen
  - HagaZiekenhuis, The Hague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arends EJ, Zlei M, Tipton CM, Cotic J, Osmani Z, de Bie FJ, Kamerling SWA, van Maurik A, Dimelow R, Gregan YI, Fox NL, Rabelink TJ, Roth DA, Sanz I, van Dongen JJM, van Kooten C, Teng YKO. Disruption of memory B-cell trafficking by belimumab in patients with systemic lupus erythematosus. Rheumatology (Oxford). 2024 Sep 1;63(9):2387-2398. doi: 10.1093/rheumatology/keae286. PMID 38775637
- [Derived] van Schaik M, Arends EJ, Soonawala D, van Ommen E, de Leeuw K, Limper M, van Paassen P, Huizinga TWJ, Toes REM, van Kooten C, Rotmans JI, Rabelink TJ, Teng YKO. Efficacy of belimumab combined with rituximab in severe systemic lupus erythematosus: study protocol for the phase 3, multicenter, randomized, open-label Synbiose 2 trial. Trials. 2022 Nov 12;23(1):939. doi: 10.1186/s13063-022-06874-w. PMID 36371234